CLINICAL TRIAL: NCT00334178
Title: A Multi-Center, Randomized, Parallel, Double-Blind, Placebo-Controlled Study in Evaluation the Efficacy and Safety of Laxymig® ER as Prophylactic Treatment in Patients With Migraine
Brief Title: Evaluation of the Efficacy and Safety of Laxymig® as Prophylactic Treatment in Patients With Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lotus Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LAXY-P001-R-2003
Record Dates: First submitted 2006-06-05; First posted 2006-06-06 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Migraine With Aura; Migraine Without Aura
Keywords: Migraine; Migraine prophylaxis
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura; Migraine Disorders | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Laxymig ER (drug)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Laxymig® ER compared with placebo in prophylactic monotherapy treatment of migraine headache.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of Laxymig® ER compared with placebo in prophylactic monotherapy treatment of migraine headache.

Four weeks baseline, following with 12 weeks treatment phase. Subjects migraine are recorded by diary cards and re-evaluated by the investigator.

Subject will have visit every 4-week (+/- 7 days).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of migraine with or without aura (typical aura with migraine headache)
* Subjects who had an average of two or more migraine frequencies per month during the 3 months before screening

Exclusion Criteria:

* Female subjects who are pregnant, lactating
* Chronic daily headache
* Previous treatment with three or more migraine prophylaxis medications failed
* Subjects with hepatic disease whose liver enzymes are over 2 times of upper limit of reference or significant dysfunction
* Coexisting medical, neurological, or psychiatric disorder that may hinder the study according to the investigator's judgment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2004-11; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
change from baseline in the frequency of migraine attacks

SECONDARY OUTCOMES:
change from baseline in 4-week in migraine periods of week 9 to 12;
change from baseline in 4-week in migraine days of week 9 to 12;
the proportion of subjects with a reduction of 50% or more in 4-week migraine frequencies;
the proportion of subjects with a reduction of 50% or more in 4-week migraine periods;
the proportion of subjects with a reduction of 50% or more in 4-week migraine days
the average symptomatic medications usage

CONTACTS AND LOCATIONS:
Overall Officials: Shuu-Jiun Wang, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (7):
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Chung-Ho Memorial Hospital, Kaohsiung Medical University, Kaohsiung City
  - Chang-Gung Memorial Hospital, Linkou District
  - Chinese Medical University Hospital, Taichung
  - SinLau Christian Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Taipei Medical University Hospital, Taipei